CLINICAL TRIAL: NCT01558713
Title: Assessment of Sensory and Motor Block After Intrathecal Administration of Bupivacaine, Ropivacaine and Levo-bupivacaine Combined With Small Doses of Fentanyl, Followed by Administration of Normal Saline Epidurally:a Clinical Trial in Parturients Scheduled for C-section
Brief Title: Epidural Volume Extension and Intrathecal Use of Local Anesthetics in Cesarean Sections
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, SKLAVOU CHRISTINA, Anesthesiologist- MD, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1312010-25
Record Dates: First submitted 2012-03-14; First posted 2012-03-20 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Stillborn Caesarean Section
Keywords: parturient
MeSH Terms: interventions — Bupivacaine; Fentanyl; Ropivacaine; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group BFS (Active Comparator): Group B: BUPIVACAINE 0,5% 2ml + 10μg FENTANYL(0,2ml) INTRATHECALLY, FOLLOWED BY EPIDURAL ADMINISTRATION OF 10 ml N/S 0,9%
  Interventions: Drug: Bupivacaine- Fentanyl - Normal Saline
- Group RFS (Active Comparator): Group R : ROPIVACAINE 0,75% 2ml + 10μg FENTANYL ( 0,2ml) INTRATHECALLY, FOLLOWED BY EPIDURAL ADMINISTRATION OF 10 ml N/S 0,9%
  Interventions: Drug: Ropivacaine-Fentanyl-Normal Saline
- Group LFS (Active Comparator): Group L: LEVO-BUPIVACAINE 0,5% 2ml + 10μg FENTANYL(0,2ml) INTRATHECALLY, FOLLOWED BY EPIDURAL ADMINISTRATION OF 10 ml N/S 0,9%
  Interventions: Drug: Levobupivacaine- Fentanyl- Normal Saline
- BupivacaineF (Active Comparator): Group BupivacaineF: BUPIVACAINE 0,5% 2ml + 10μg FENTANYL(0,2ml) INTRATHECALLY
  Interventions: Drug: Bupivacaine + Fentanyl
- RopivacaineF (Active Comparator): Group RopivacaineF : ROPIVACAINE 0,75% 2ml + 10μg FENTANYL ( 0,2ml) INTRATHECALLY.
  Interventions: Drug: Ropivacaine + Fentanyl
- LevobupivacaineF (Active Comparator): Group LevobupivacaineF: LEVO-BUPIVACAINE 0,5% (2ml) + 10μg FENTANYL(0,2ml) INTRATHECALLY.
  Interventions: Drug: Levobupivacaine + Fentanyl

INTERVENTIONS:
Drug: Bupivacaine- Fentanyl - Normal Saline — Bupivacaine 0,5%, 2ml (10mg)bolus, Fentanyl 50μg/ml, 0,2ml (10 μg)bolus, Normal Saline 0,9%, 10ml bolus
  Other Names: Bupivacaine hydrochloride 0.5% ( Marcaine Spinal, 5 mg/ml, AstraZeneca, Missisipi, ON, Canada); Fentanyl, 50μg/ml, Janssen-Cilag, Belgium; 0,9% Sodium Chloride Inj. BP, B.BRAUN Melsungen AG, German
  Arms: Group BFS
Drug: Ropivacaine-Fentanyl-Normal Saline — Ropivacaine 0,75%, 2ml (15mg)bolus, Fentanyl 50μg/ml, 0,2ml (10 μg)bolus, Normal Saline 0,9%, 10ml bolus
  Other Names: Ropivacaine 0.75% :( Naropeine 7.5mg/ml, AstraZeneca); Fentanyl: 50μg/ml, Janssen-Cilag, Belgium; 0,9% Sodium Chloride Inj. BP, B.Braun Melsungen AG
  Arms: Group RFS
Drug: Levobupivacaine- Fentanyl- Normal Saline — Levo-bupivacaine 0,5%, 2ml (10mg)bolus, Fentanyl 50μg/ml, 0,2ml (10 μg)bolus, Normal Saline 0,9%, 10ml bolus
  Other Names: Chirocaine 5mg/ml, Abbot Laboratories, Greece; Fentanyl, 50μg/ml, Janssen-Cilag, Belgium; 0,9% Sodium Chloride Inj. BP, B.Braun Melsungen AG
  Arms: Group LFS
Drug: Bupivacaine + Fentanyl — Bupivacaine 0,5%, 2ml (10mg)bolus, Fentanyl 50μg/ml, 0,2ml (10 μg)bolus
  Other Names: Bupivacaine hydrochloride 0,5% (Marcaine Spinal, 5mg/ml,AstraZeneca,Missisipi, ON, Canada); Fentanyl, 50μg/ml (Janssen-Cilag, Belgium)
  Arms: BupivacaineF
Drug: Ropivacaine + Fentanyl — Ropivacaine 0,75%, 2ml (15mg)bolus, Fentanyl 50μg/ml, 0,2ml (10 μg)bolus.
  Other Names: Ropivacaine 0,75% :(Naropeine 7,5mg/ml, AstraZeneca); Fentanyl 50μg/ml, Janssen-Cilag, Belgium.
  Arms: RopivacaineF
Drug: Levobupivacaine + Fentanyl — Levo-bupivacaine 0,5%, 2ml (10mg)bolus, Fentanyl 50μg/ml, 0,2ml (10 μg)bolus
  Other Names: Chirocaine 5mg/ml, Abbot Laboratories, Greece.; Fentanyl 50μg/ml, Janssen-Cilag, Belgium.
  Arms: LevobupivacaineF

SUMMARY:
Intrathecal (i.t.) administration of isobaric bupivacaine, ropivacaine and levobupivacaine with addition of fentanyl for c-section either combined or not with administration of 10 ml of N/S 0,9% epidurally, in order to extent epidural space.Sensory and motor block profile, haemodynamics and side effects were assessed.

DETAILED DESCRIPTION:
Parturients scheduled for elective caesarean section are randomly allocated to 6 groups: they receive double-blindly intrathecal isobaric bupivacaine 10 mg ( Group B), ropivacaine 15mg (Group R) , levobupivacaine 10mg (Group L) combined with 10 μg fentanyl and followed by epidural administration of 10 ml of N/S 0,9% respectively, and isobaric bupivacaine 10 mg ( Group BupivacaineF), ropivacaine 15mg (Group RopivacaineF) , and levobupivacaine 10mg (Group LevobupivacaineF) combined with 10 μg fentanyl without epidural administration of 10 ml of N/S 0,9%. Clinical endpoints are the sensory and motor block profile, haemodynamics (arterial pressure, heart rate) and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean section
* ASA I-II

Exclusion Criteria:

* complicated pregnancy (i.e preeclampsia, eclampsia,arterial hypertension, diabetes mellitus)
* abnormal fetal heart rate at the time of admission
* body mass index > 35 kg/m2
* height <150cm and >185 cm
* age <18 yrs and >40 yrs
* patients with contraindication to spinal anaesthesia( i.e anticoagulants)
* ASA >III
* intraoperative excessive bleeding
* patients with previous psychiatric diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Dermatomes of Sensory block | up to 120 minutes average
  Dermatomes of sensory block(pin prick test) are assessed every minute for the first 30 minutes after the intrathecal administration of local anesthetics and there after every 5 minutes until withdrawal of sensory block
Motor block | up to 120 minutes average
  Motor block according to the Bromage scale are assessed every minute for the first 30 minutes after the intrathecal administration of local anesthetics and there after every 5 minutes until withdrawal motor block

SECONDARY OUTCOMES:
Arterial Blood Pressure | up to 120 minutes average
  Measurements assesed every minute within the first 30 minutes after the intrathecal administration of local anesthetics and every 5 minutes until withdrawal of sensory and motor block

CONTACTS AND LOCATIONS:
Overall Officials: KRITON S FILOS, PROFESSOR, Study Chair — Department of Anesthesiology and Intensive Care Medicine, University Hospital of Patras; Christina G Sklavou, MD, Principal Investigator — Department of Anesthesia and Intensive Care Medicine, University Hospital of Patras
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, University Hospital of Patras, Pátrai, Achaia, Greece